CLINICAL TRIAL: NCT04923074
Title: the Application of Diffusion Tensor Imaging(DTI) in the Evaluation of Peripheral Neuropathy in Anti-neutrophil Cytoplasmic Antibodies Associated Vasculitis(AAV)
Brief Title: the Application of Diffusion Tensor Imaging in the Evaluation of Peripheral Neuropathy in ANCA Associated Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-162
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: ANCA Associated Vasculitis
Keywords: peripheral neuropathy
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DTI group: the patient in this group will receive DTI evaluation
  Interventions: Other: diffusion tensor imaging(DTI) evaluation
- routine group: the patient in this group will receive routine evaluation

INTERVENTIONS:
Other: diffusion tensor imaging(DTI) evaluation — DTI is a new kind of MRI technique to evaluate peripheral neuropathy
  Groups: DTI group

SUMMARY:
1. Include qualified 50 ANCA-associated vasculitis(AAV) patients; and the first 27 patients will be divided into 3 groups with different diffused tension image (DTI) parameters and to choose the best strategy；
2. On baseline, 6 months after treatment and 24 months after treatment, the AAV patients will accomplish the Birming-ham vasculitis activity score(BVAS) besides DTI；
3. The new serum biomarkers of AAV associated peripheral neuropathy will be measured by ELISA； (4) Another cohort with 50 patients with AAV associated peripheral neuropathy who were evaluated by traditional methods (electromyogram) and compared to the patients cohort that evaluated using DTI by cost-benefit analysis

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80 years old；
* must fulfill 2012 criteria of ANCA associated vasculitis
* presented with peripheral neuropathy diagnosed by specialists

Exclusion Criteria:

* the ANCA associated vasculitis is already in the stable stage after treatments
* any vital organ dysfunction
* active infection or cancer
* can not finish DTI scan

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult AAV patients with peripheral neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
To assess the optimal b-value (a key parameter) for DTI in AAV associated peripheral neuropathy | 2 years
  b-value is a key technique parameter for DTI, which will decide the quality of DTI image

SECONDARY OUTCOMES:
the association between normative diffusion value of DTI (FA and ADC value) and disease activity activity score of AAV (BVAS). | 2 years
  Birmingham Vasculitis Activity Score (BVAS) is a index of vasculitis disease activity, with the score range 0-63. Fractional anisotropy(FA) and apparent diffusion coefficient(ADC) are two parameters that can be read through DTI image .
the association between normative diffusion value of DTI (FA and ADC value) and serum biomarkers of AAV associated neuropathy | 2 years
  sCD163, Nfl（neurofilament light polypeptide）and OPN（osteopontin）are new biomarkers of peripheral neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xue, Study Chair — 2nd affiliated hospital of Zhejiang University, School of Medicine
Locations (1):
- 2nd affiliated hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China